CLINICAL TRIAL: NCT03991156
Title: AVATAR Anesthesia Alternative in Pediatric Radiotherapy: A Multi-Center Study
Status: Active, not recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-47864; PEDSVAR0050 (Other: OnCore); IRB-47864 (Other: Stanford IRB)
Record Dates: First submitted 2019-06-12; First posted 2019-06-19 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia
Keywords: Radiotherapy
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Audio-Visual Assisted Therapeutic Ambience in Radiotherapy
  Interventions: Device: Audio-Visual Assisted Therapeutic Ambience in Radiotherapy; Other: Quality of Life Survey, PedsQL3.0; Other: Yale Preoperative Anxiety Scale Short Form (mYPAS-SF)

INTERVENTIONS:
Device: Audio-Visual Assisted Therapeutic Ambience in Radiotherapy — Audio Visual System
  Other Names: AVATAR
Other: Quality of Life Survey, PedsQL3.0 — Quality of life survey using the PedsQL 3.0 Cancer Module
Other: Yale Preoperative Anxiety Scale Short Form (mYPAS-SF) — Yale Preoperative Anxiety Scale Short Form (mYPAS-SF).[24] is a survey to measure anxiety

SUMMARY:
To determine the success rate of the AVATAR audio-visual system. All patients enrolled in the study will be counted, and each patient who is able to undergo at least one fraction without anesthesia will count as a success while each patient who does not have at least one fraction without anesthesia will count as a failure. The success rate will be the proportion of patients who are successes.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients ages 3-10 receiving radiotherapy qualify for enrollment.
* The patient must speak English or Spanish.

Exclusion Criteria:

* If parent/guardian is unable to take part in helping to complete questionnaires
* Patients with malignancies of the eye for which radiation is planned
* Patients that do not speak English or Spanish

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The age range of patients is 3-10 years old, and there is no discrimination on ethnic background in recruitment for this study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Success rate of AVATAR system | 24 months
  Success rate will be determined as the proportion of patients who are successes.
  Success will be counted as each patient who is able to undergo at least one fraction without anesthesia while each patient who does not have at least one fraction without anesthesia will count as a failure.

SECONDARY OUTCOMES:
Measure Fractional Success using AVATAR system | 24 months
  Fractional Success will be is counted as a fraction in which the patient does not require anesthesia will count as a fractional success, while a fraction in which the patient required anesthesia will be a fractional failure.
Determine the difference in patient anxiety between successful AVATAR patients and not-successful patients. | 24 months
  The difference in patient anxiety between successful AVATAR patients and not-successful patients will be determined. Anxiety will be assesed by modified Yale Preoperative Anxiety Survey Short Form (mYPAS-SF). mYPAS-SF measurement instrument uses 5 items, each representing a different domain of child anxiety, and is used at 4 points in time.
Compare the rates of anesthesia with historical controls | 24 months
  Compare the rates of anesthesia use between patients using AVATAR to historical controls who were not introduced to AVATAR.
Determine the rate at which patients convert from requiring anesthesia to not requiring anesthesia while using AVATAR | 24 months
  The rate at which patients convert from requiring anesthesia to not requiring anesthesia while using AVATAR will be determined. Conversion is determined by the fraction at which the patient switches from using anesthesia to not using anesthesia.
Difference in health quality of life between subjects with or without anesthesia | 24 months
  The difference between family-reported health-related quality of life between patients who were able to tolerate treatment without anesthesia using the AVATAR program and patients who required anesthesia for the entire treatment. The quality of life will be measured using Pediatric oncology quality of life inventory 3.0-cancer module (PedsQL 3.0 Cancer Module)
Assess predictability for AVATAR patient success | 24 months
  AVATAR patient success will be determined by using the predictability of the PedsQL3.0 Cancer and modified Yale Preoperative Assessment Survey Short Form (mYPAS-SF) questionnaires. mYPAS-SF measurement instrument uses 5 items, each representing a different domain of child anxiety, and is used at 4 points in time.

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Hiniker, Principal Investigator — Stanford University
Locations (11):
- United States (11):
  - Stanford University, Stanford, California
  - Indiana University, Bloomington, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute/Brigham & Women Children Hospital, Boston, Massachusetts
  - University of Minnesota, Minneota, Minnesota
  - St. Louis Children's Hospital, St Louis, Missouri
  - University of Rochester School of Medicine, Rochester, New York
  - University North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's/UC Health Proton Therapy Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - St. Jude Children Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gutkin PM, Skinner L, Jiang A, Donaldson SS, Loo BW Jr, Oh J, Wang YP, von Eyben R, Snyder J, Bredfeldt JS, Breneman JC, Constine LS, Faught AM, Haas-Kogan D, Holmes JA, Krasin M, Larkin C, Marcus KJ, Maxim PG, McClelland S 3rd, Murphy B, Palmer JD, Perkins SM, Shen CJ, Terezakis S, Bush K, Hiniker SM. Feasibility of the Audio-Visual Assisted Therapeutic Ambience in Radiotherapy (AVATAR) System for Anesthesia Avoidance in Pediatric Patients: A Multicenter Trial. Int J Radiat Oncol Biol Phys. 2023 Sep 1;117(1):96-104. doi: 10.1016/j.ijrobp.2023.03.063. Epub 2023 Mar 30. PMID 37001762